CLINICAL TRIAL: NCT03633656
Title: Iron Dosing Pilot Study Using Model Predictive Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Alfred Jacobs, Assoc Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: KDP001 IRB#18.0761
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Renal Insufficiency, Chronic; Anemia, Iron Deficiency; Anemia of Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Model predictive control recommendation of iron dosing in combination with an erythropoietic stimulating agent.
  Interventions: Device: Model predictive control; Device: Model Predictive Control of Iron Dosing

INTERVENTIONS:
Device: Model predictive control — Computer aided dose selection for the treatment of iron deficient anemia.
Device: Model Predictive Control of Iron Dosing — Model Predictive Control of Iron Dosing

SUMMARY:
This is a pilot study to test the utility of an integrated approach in the management of the anemia of chronic kidney disease through the administration of both an erythropoietic stimulating agent and iron. Subjects will be studied for 6 months during which all iron dosing will be recommended using a computer based tool using model predictive control. Comparisons will be made to the 6 months prior to enrollment in to the study.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease
* anemia
* receiving intravenous iron

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of tsat values within range | Monthly for 6 months
  Tsat is measured as a percent saturation, desired range is 20 to 50%

SECONDARY OUTCOMES:
Iron dose over ride by physician | Monthly for 6 months
  Number of recommended iron doses that the prescribing physician altered.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Jacobs, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No